CLINICAL TRIAL: NCT04784286
Title: Telemedicine Follow-up for Bariatric Surgery Patients: What Do Patients Prefer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of Covid-19, in-person visits were halted and telemedicine was used.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elizabeth B. Habermann, Professor of Health Services Research, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 18-010144
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Care Provider, Investigator
Masking Description: The randomized assignments (2 arms) will be generated by an analyst/statistician using a Mayo Clinic statistical application. The research assistant/coordinator will issue the next in a series of sequentially numbered, sealed, opaque envelopes containing the group assignment. The envelope will have information regarding the treatment assignment and will be entered into a database by the study coordinator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine 30-day follow-up visit (Active Comparator): The Center for Connected Care will arrange for 30-day post-op telemedicine visits via a secured video application. When there is a telemedicine visit, the Center of Connected Care will connect the patient and then page the midlevel provider and dietitian after the electronic rooming process is complete & the patient is ready.
  A survey about post-operative care visits within 7-14 days after that visit. The survey will focus on the following aspects: baseline familiarity with technology, patients' satisfaction with the post-op care they received, patients' preference of in-person vs telemedicine visits, patients' estimation of additional costs for care outside of the direct medical costs, along with an open question asking for comments & feedback about their overall experience with their follow-up appointment.
  Interventions: Other: Telemedicine 30-day post-op visit
- In-person 30-day follow-up visit (Active Comparator): Standard practice of having bariatric surgery patients follow up with the bariatric surgery midlevel providers as well as with dietitians within 30-days after their bariatric procedure. The bariatric surgery midlevel providers are staffed and supported by our bariatric surgeons in case if they have questions or concerns.
  Participants will be contacted via telephone and will be surveyed about their post-operative care visits within 7-14 days after that visit. The survey will focus on the following aspects: baseline familiarity with technology, patients' satisfaction with the post-operative care they received, patients' preference of in-person vs telemedicine visits, patients' estimation of additional costs for their care outside of the direct medical costs, along with an open question that will ask patients to provide comments and feedback about their overall experience with their follow-up appointment.
  Interventions: Other: In-Person 30-day post-op visit

INTERVENTIONS:
Other: Telemedicine 30-day post-op visit — Consented subjects randomized to the telemedicine visit arm will do their 30-day post-op visit via secure telemedicine video application through the Center of Connected Care. A survey will be asked via telephone about their post-op care visit, costs incurred, and feedback.
  Other Names: Patient Satisfaction
  Arms: Telemedicine 30-day follow-up visit
Other: In-Person 30-day post-op visit — Consented subjects randomized to the in-person visit arm will physically come to a clinical visit with the bariatric surgery midlevel providers. A survey will be asked via telephone about their post-op care visit, costs incurred, and feedback.
  Other Names: Patient Satisfaction
  Arms: In-person 30-day follow-up visit

SUMMARY:
This is a randomized clinical trial that will randomize bariatric patients undergoing laparoscopic sleeve gastrectomy or laparoscopic Roux-en-Y gastric bypass to receive either in-person or telemedicine post-operative follow-up within 30 days after surgery.

DETAILED DESCRIPTION:
Our current bariatric practice: Bariatric surgery patients are expected to follow up with the bariatric surgery midlevel providers as well as with dietitians within 30-days after their bariatric procedure. The bariatric surgery midlevel providers are staffed and supported by our bariatric surgeons in case if they have questions or concerns. Patients do not get billed for post-operative visits within 90-days of global surgery period; the same global surgery rules apply to both in-person and telemedicine visits.

Patients are required to follow-up after surgery as part of the Metabolic and Bariatric Surgery Accreditation and Quality Improvement Program.

Adult (≥ 18 year-old) participants in the study will undergo primary Roux-en Y gastric bypass or sleeve gastrectomy and will randomized to telemedicine or in-person visit before their surgical procedure.

Patients who encounter unexpected intra-operative or post-operative complication or unexpected hospital course may not be offered telemedicine visits but will be included in our analysis. The performing surgeon will determine if a patient is illegible for telemedicine visit if unexpected course was encountered. However, analysis will be analysis to treat.

All participants will be contacted via telephone and will be surveyed about their post-operative care visits within 7-14 days after that visit, which is typically performed within 30-days after surgery. The survey will be developed in coordination with the Mayo Clinic Research Survey Center and will focus on the following aspects: baseline familiarity with technology, patients' satisfaction with the post-operative care they received, patients' preference of in-person vs telemedicine visits, patients' estimation of additional costs for their care outside of the direct medical costs, along with an open question that will ask patients to provide comments and feedback about their overall experience with their follow-up appointment.

ELIGIBILITY:
Inclusion Criteria:

Patients > 18 years of age Having bariatric surgery; primary Roux-en Y gastric bypass or sleeve gastrectomy Be in the United States at the time of their 30-day follow-up Live 70 miles or further from Mayo Clinic downtown campus in Rochester, MN Access to WI-FI and electronic device (laptop, computer, tablet, smart phone, etc.) Willing to consent for the study

Exclusion Criteria:

Patients < 18 years of age Be outside the United States at the time of their follow-up Undergoing revision of previous bariatric surgery Unable to speak English Unwilling or unable to provide consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Patients' preference of telemedicine or in-person assessment for post-operative care. | 30 day post-op
  This will be addressed by asking the following question in the survey:
  How likely or unlikely would you be to accept an invitation to meet with your bariatric provider via video call from your home when you do not need new labs/imaging, your physician can review outside labs/imaging, and no physical exam/procedure is needed?

SECONDARY OUTCOMES:
Post-operative complication rates are similar between patients receiving telemedicine and standard post-operative clinic visits. | 30 day post-op
  Complication rates in both groups including unplanned readmission or re-operation
Patients' out-of-pocket costs for attending telemedicine post-operative visits are less than attending standard clinic. | 30 day post-op
  Patients' estimated out-of-pocket costs of follow-up visits, including missed days of work, hotel stays and transportation
Institutional costs needed to provide telemedicine visits are less than what is needed for standard clinic care. | 30 day post-op
  Compare institutional costs needed to provide telemedicine with those to provide standard post-operative care for bariatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Habermann, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
All individual participant data will be deidentified by giving each consented subject a unique number/code before sharing with the other researchers.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials